CLINICAL TRIAL: NCT06093191
Title: Efficacy and Safety of tobRamycin Inhalation Solution for Pseudomonas AeruginoSa Eradication in Bronchiectasis (ERASE): a Multi-center, 2×2 Factorial Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Tobramycin Inhalation Solution for Pseudomonas Aeruginosa Eradication in Bronchiectasis
Acronym: ERASE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20230329
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Bronchiectasis Adult; Pseudomonas Aeruginosa Infection
Keywords: bronchiectasis,; Pseudomonas Aeruginosa; eradication; inhaled antibiotics; randomized controlled trial
MeSH Terms: conditions — Pseudomonas Infections; Bronchiectasis | interventions — Ciprofloxacin; Anti-Bacterial Agents

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into one of the four groups. No cross-over of the study group will be made
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both investigators and participants were blinded to the treatment assignment throughout the study. To maintain this blinding, placebos were used, which were made indistinguishable in appearance from the inhaled tobramycin solution and oral ciprofloxacin. The taste of the inhaled tobramycin solution was not disclosed to the patients, and neither the patients nor most clinicians had prior knowledge of its taste. This blinding approach ensures that both participants and investigators remain unaware of the specific treatment each patient is receiving, thereby reducing potential biases in the study's results
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Combination group (Active Comparator): Participants will receive inhaled 300mg of tobramycin solution twice daily for 12 weeks and oral 750mg of ciprofloxacin twice daily for 2 weeks
  Interventions: Drug: Tobramycin Inhalant Product; Drug: Ciprofloxacin 750 MG
- Tobramycin inhalation solution alone group (Active Comparator): Participants will receive inhaled 300mg of tobramycin twice daily for 12 weeks and oral ciprofloxacin placebo twice daily for 2 weeks
  Interventions: Drug: Tobramycin Inhalant Product; Drug: Oral ciprofloxacin placebo
- Oral ciprofloxacin alone group (Active Comparator): Participants will receive oral 750mg of ciprofloxacin twice daily for 2 weeks and inhaled saline twice daily for 12 weeks
  Interventions: Drug: Ciprofloxacin 750 MG; Drug: Natural saline inhalation
- Placebo group (Placebo Comparator): Participants will receive inhaled saline twice daily for 12 weeks and oral ciprofloxacin placebo twice daily for 2 weeks
  Interventions: Drug: Oral ciprofloxacin placebo; Drug: Natural saline inhalation

INTERVENTIONS:
Drug: Tobramycin Inhalant Product — Tobramycin will be nebulized (300mg twice daily) with an ultrasonic nebulizer. A total of 12 weeks therapy will be scheduled.
  Other Names: Inhaled antibiotics
  Arms: Combination group; Tobramycin inhalation solution alone group
Drug: Ciprofloxacin 750 MG — Oral ciprofloxacin 750mg twice daily will be prescribed for 2 weeks.
  Other Names: Oral antibiotics
  Arms: Combination group; Oral ciprofloxacin alone group
Drug: Oral ciprofloxacin placebo — Oral ciprofloxacin placebo twice daily will be prescribed for 2 weeks.
  Other Names: Oral antibiotics
  Arms: Placebo group; Tobramycin inhalation solution alone group
Drug: Natural saline inhalation — Natural saline will be nebulized (5ml twice daily) with an ultrasonic nebulizer. A total of 12 weeks therapy will be scheduled.
  Other Names: Inhaled saline
  Arms: Oral ciprofloxacin alone group; Placebo group

SUMMARY:
People with bronchiectasis are prone to Pseudomonas aeruginosa (PA) infections, which can become chronic and lead to increased death rates and disease severity. Studies from cystic fibrosis suggest that eradication therapy aimed at PA can successfully transition patients to a culture-negative status, providing long-term benefits. Current guidelines for managing bronchiectasis in adults recommend eradicating PA when it is first or newly isolated; however, there is a lack of randomized controlled trials supporting such recommendations. The researchers hypothesize that both oral ciprofloxacin combined with Tobramycin inhalation solution and Tobramycin inhalation solution alone are superior to no eradication (inhaled saline) in terms of the eradication rates of PA, defined as a negative sputum culture of PA at both 24 weeks and 36 weeks.

DETAILED DESCRIPTION:
The presence of Pseudomonas aeruginosa (PA) in bronchiectasis patients is associated with a greater impairment in lung function, increased systemic and airway inflammation, more frequent exacerbations, decreased quality of life, a higher risk of hospitalization, and increased mortality. Current guidelines recommend eradicating PA when it is first isolated, but there is limited randomized controlled trial evidence to support this.

In cystic fibrosis, early infection with PA is clearly linked to worse outcomes, and eradication is associated with clinical benefits, including improved lung function and reduced hospitalization. Small sample observational studies have shown that eradication therapy following initial PA isolation is efficient, with eradication rates of 40%-57% in bronchiectasis. Therefore, a randomized control trial of PA eradication therapy is needed to determine the microbiological and clinical outcomes of this therapy.

There is also uncertainty about whether inhaled antibiotics alone are sufficient to eradicate PA in non-cystic fibrosis bronchiectasis, given the less severe nature of the disease compared to cystic fibrosis. It's unclear whether adding another antibiotic, such as oral ciprofloxacin in this study, to inhaled antibiotics at the initial stage is necessary as an enhanced treatment for eradicating PA in bronchiectasis.

To address these knowledge gaps, a multicenter, 2×2 factorial randomized, double-blind, placebo-controlled, parallel-group study is designed in bronchiectasis patients with newly or firstly isolated PA. This study aims to investigate the efficacy and safety of tobramycin inhalation solution alone or in combination with oral ciprofloxacin in eradicating PA in bronchiectasis.

Patients will be randomly assigned to one of four groups:

1. Placebo group: participants will receive inhaled saline twice daily for 12 weeks and an oral ciprofloxacin placebo twice daily for 2 weeks.
2. Oral ciprofloxacin alone group: participants will receive 750mg of oral ciprofloxacin twice daily for 2 weeks and inhaled saline twice daily for 12 weeks.
3. Tobramycin inhalation solution alone group: participants will receive 300mg of inhaled tobramycin twice daily for 12 weeks and an oral ciprofloxacin placebo twice daily for 2 weeks.
4. Combination group: participants will receive 300mg of inhaled tobramycin solution twice daily for 12 weeks and 750mg of oral ciprofloxacin twice daily for 2 weeks.

This study will provide valuable insights into the most effective treatment strategy for eradicating PA in bronchiectasis patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 years and 80 years at screening
2. Signed and dated written informed consent prior to admission to the study in accordance with local legislation.
3. Clinical history consistent with bronchiectasis (cough, chronic sputum production and/or recurrent respiratory infections) and investigator-confirmed diagnosis of bronchiectasis by CT scan
4. During the screening period, patients must have a positive P. aeruginosa culture in their sputum and must meet one of the following criteria: (1) they have never been isolated with P. aeruginosa from sputum or bronchoalveolar lavage fluid (BALF) before; (2) they were isolated with P. aeruginosa from sputum or BALF for the first time within 12 months before screening; (3) they had prior isolation of P. aeruginosa but not within the last 24 months (defined as having negative sputum culture results at least twice before starting antibiotic treatment)
5. During the screening period, patients must remain clinically stable (no significant changes in respiratory symptoms and no upper respiratory tract infection or bronchiectasis exacerbations for 4 weeks)
6. During the screening period, P. aeruginosa is not resistant to Tobramycin and Ciprofloxacin based on the drug sensitivity test of sputum culture in vitro
7. Patient can tolerate nebulized inhalation therapy

Exclusion criteria

1. Patients who are allergic to or cannot tolerate the investigational drugs (Tobramycin, Ciprofloxacin)
2. Patients with uncontrolled asthma, physician-diagnosed cystic fibrosis, and Current diagnosis of allergic bronchopulmonary aspergillosis, hypogammaglobulinemia, common variable immunodeficiency, mycobacterial infection (including pulmonary non-tuberculous mycobacterial disease) requiring treatment.
3. Participants with unstable cardiovascular and cerebrovascular diseases, defined as those who have experienced clinically worsening symptoms (such as unstable angina, rapid atrial fibrillation, cerebral hemorrhage, acute cerebral infarction, etc.) or have been hospitalized due to these diseases within 90 days prior to the screening
4. Participants with progressive or uncontrolled systemic diseases, such as those affecting the urinary, hematological, digestive, endocrine, respiratory, circulatory, nervous, or mental systems, are not suitable for this clinical trial. This is particularly the case if these conditions are evaluated by the researcher as being unstable or potentially escalating into severe conditions during the trial.
5. AST and/or ALT >2 ULN at screening period
6. Serum creatinine >ULN at screening period
7. Participants with a history of hearing loss or those who are determined by the researcher to have clinically significant chronic tinnitus
8. Participants with a history of prolonged QT intervals or those whose electrocardiograms show prolonged QT intervals during the screening period
9. Participants who have used drugs that are prohibited according to the plan during the screening period.
10. Women of childbearing potential adhering to contraception requirements.
11. Patients with FEV1% of predicted value<30%
12. Participants who have participated in other clinical trials (defined as those where medication has been administered) within the 4 weeks prior to the screening
13. Participants who have experienced moderate or severe hemoptysis (defined as expectorating 100-500ml of blood in 24 hours for moderate hemoptysis; and expectorating more than 500ml in 24 hours, or a single instance of expectorating more than 100ml of blood for severe hemoptysis) due to bronchiectasis within the past 6 months.
14. Participants who are deemed unsuitable for inclusion in the study due to other reasons, as determined by the researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients successfully eradicating PA in each group by the end of the study, defined as a negative sputum culture of PA at both 24 weeks and 36 weeks. | 36 weeks
  The proportion of patients with negative PA from sputum samples, either spontaneous or induced, in each group by the end of the study, at both 24 and 36 weeks post-randomization

SECONDARY OUTCOMES:
The proportion of patients in each group who have a negative Pseudomonas aeruginosa (PA) culture 12 weeks after randomization | 12 weeks
  The proportion of patients in each group who have a negative Pseudomonas aeruginosa (PA) culture 12 weeks after randomization
The proportion of patients in each group who have a negative Pseudomonas aeruginosa (PA) culture 24 weeks after randomization | 24 weeks
  The proportion of patients in each group who have a negative Pseudomonas aeruginosa (PA) culture 24 weeks after randomization
The proportion of patients in each group who have a negative Pseudomonas aeruginosa (PA) culture 36 weeks after randomization | 36 weeks
  The proportion of patients in each group who have a negative Pseudomonas aeruginosa (PA) culture 36 weeks after randomization
Time to the first bronchiectasis exacerbation since randomization | 36 weeks
  Time to the first bronchiectasis exacerbation since randomization
Frequency of bronchiectasis exacerbation since randomization | 36 weeks
  Frequency of bronchiectasis exacerbation since randomization
Frequency of bronchiectasis exacerbation since randomization | 12 weeks
  Frequency of bronchiectasis exacerbation since randomization
Frequency of hospitalization due to bronchiectasis exacerbation since randomization | 36 weeks
  Frequency of hospitalization due to bronchiectasis exacerbation since randomization
Frequency of hospitalization due to bronchiectasis exacerbation since randomization | 12 weeks
  Frequency of hospitalization due to bronchiectasis exacerbation since randomization
Time to reoccurrence of P. aeruginosa infection since randomization | 36 weeks
  Time to reoccurrence of P. aeruginosa infection since randomization
Quality-of-Life-Bronchiectasis Respiratory Symptom Scale, that measures health-related quality of life | Assessed at baseline, 12 weeks, 24 weeks and 36 weeks post-randomization.
  The Quality-of-Life-Bronchiectasis (QoL-B) questionnaire is a disease-specific survey designed for patients with bronchiectasis. The Respiratory Symptoms scale is a component of the QoL-B questionnaire, with a scale range from 0 to 100. Higher scores on this scale signify a better health status.
St.George Respiratory Questionnaire, that measures health-related quality of life | Assessed at baseline, 12 weeks, 24 weeks and 36 weeks post-randomization.
  St.George Respiratory Questionnaire (SGRQ): a validated questionnaire for use in bronchiectasis population. This questionnaire is structured into 3 main components: symptoms, activity and impacts.
  Scale range is 0-100, where lower scores correspond to the better health status.
  Each questionnaire response has a unique empirically derived "weight".
  Each component of the questionnaire is scored separately in three steps:
  i. The weights for all items with a positive responses are summed. ii. The weights for missed items are deducted from the maximum possible weight for each component. The weights for all missed items are deducted from the maximum possible weight for the Total score.
  iii. The score is calculated by dividing the summed weights by the adjusted maximum possible weight for that component and expressing the result as a percentage The Total score is calculated in similar way.
Euroqual-5 Dimensions questionnaire | Assessed at baseline, 12 weeks, 24 weeks and 36 weeks post-randomization.
  The Euroqual-5 Dimensions questionnaire (EQ-5D) consists of two parts: health state description and evaluation. In the description part, health status is measured across five dimensions (5D): mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Respondents rate their severity level for each dimension using a five-level (EQ-5D-5L) scale.
  In the evaluation part, respondents assess their overall health status using the visual analogue scale (EQ-VAS), which ranges from 0 to 100, with higher scores indicating a better health status.
  Health states defined by the EQ-5D-5L descriptive system are converted into index values. This facilitates the calculation of Quality-Adjusted Life Years (QALYs), which are used to inform economic evaluations of healthcare interventions, according to guidelines found at https://euroqol.org.
Changes in forced expiratory volume in 1 second [FEV1] at 12, 24, and 36 weeks compared with baseline | Assessed at baseline, 12 weeks, 24 weeks and 36 weeks post-randomization.
  Changes in forced expiratory volume in 1 second [FEV1] at 12, 24, and 36 weeks compared with baseline
Changes in forced vital capacity [FVC] at 12, 24, and 36 weeks compared with baseline | Assessed at baseline, 12 weeks, 24 weeks and 36 weeks post-randomization.
  Changes in forced vital capacity [FVC] at 12, 24, and 36 weeks compared with baseline
Changes in forced expiratory flow at 25-75% of forced vital capacity at 12, 24, and 36 weeks compared with baseline | Assessed at baseline, 12 weeks, 24 weeks and 36 weeks post-randomization.
  Changes in forced expiratory flow at 25-75% of forced vital capacity at 12, 24, and 36 weeks compared with baseline
The cost of hospitalization | 36 weeks
  The cost of hospitalization during the whole study period
Other sputum microbiology during the whole study period. | 36 weeks
  Sputum cultures were conducted at baseline, 2 weeks, 8 weeks, 12 weeks, 24 weeks, and 36 weeks. Other sputum microbiology, including Staphylococcus aureus, Escherichia coli, Klebsiella pneumoniae, Streptococcus pneumoniae, Haemophilus influenzae, Moraxella catarrhalis, Burkholderia cepacia complex, Stenotrophomonas, Aspergillus, and Candida spp. were documented throughout the entire study period. The number of participants who yielded at least one positive culture for these microorganisms was calculated.
Resistant P. aeruginosa during the whole study period | 36 weeks
  Sputum cultures were performed at intervals of 2 weeks, 8 weeks, 12 weeks, 24 weeks, and 36 weeks. Drug sensitivity testing was conducted to assess the resistance of the current P. aeruginosa sample to antibiotics such as ciprofloxacin and tobramycin. The number of participants who showed growth of Pseudomonas aeruginosa resistant to ciprofloxacin and/or tobramycin was calculated.
Number of adverse events | 36 weeks
  Reported by the PI or designee via interview with patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Fu Xu, PhD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (63):
- China (63):
  - Hainan General Hospital, Hainan Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Qilu Hospital of Shandong University, Jinan, Shangdong
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - The Shanghai Fifth People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai pulmonary hospital, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang
  - The First People's Hospital of Anning City Affiliated to Kunming University of Science and Technology, Anning
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing
  - Peking University Third Hospital, Beijing
  - The First Affiliated Hospital of Jilin University, Changchun
  - The Second Xiangya Hospital of Central South University, Changsha
  - Xiangya Hospital, Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - The Third Affiliated Hospital of Chongqing Medical University, Chongqing
  - The Second Affiliated Hospital of Dalian Medical University, Dalian
  - Fujian Provincial Hospital, Fuzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine, Guangzhou
  - Guizhou Provincial People's Hospital, Guiyang
  - The Second Affiliated Hospital of Zhengjiang University, Hangzhou
  - Anhui Chest Hospital, Hefei
  - The First Affiliated Hospital of Anhui Medical University, Hefei
  - Huzhou Central Hospital, Huzhou
  - The First Hospital of Jiaxing City, Jiaxing
  - The Second Hospital of Jiaxing City, Jiaxing
  - The First Affiliated Hospital of Shandong First Medical University, Jinan
  - The First Affiliated Hospital of Wenzhou Medical University, Jinan
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Affiliated Sir Run Run Hospital of Nanjing Medical University, Nanjing
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Affiliated Hospital, Nantong University, Nantong
  - The Sixth People's Hospital of Nantong City, Nantong
  - Fenghua District People's Hospital of Ningbo City, Ningbo
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - The First Affiliated Hospital of Ningbo University, Ningbo
  - Qingdao Municipal Hospital, Qingdao
  - Baoshan District Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai
  - Shanghai Eighth People's Hospital, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shanghai Putuo District People's Hospital, Shanghai
  - Shanghai Shidong Hospital of Yangpu District, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai
  - Shanghai Songjiang District Central Hospital, Shanghai
  - Shanghai Yangpu District Central Hospital, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai
  - Shangrao People's Hospital, Shangrao
  - Shengjing Hospital of China Medical University, Shenyang
  - The First Affiliated Hospital of China Medical University, Shenyang
  - Shenzhen Institute of Respiratory Diseases, Shenzhen
  - The Eighth Affiliated Hospital of Sun Yat-Sen University, Shenzhen
  - Suzhou Science and Technology Town Hospital, Suzhou
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Union Hospital,Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Subei People's Hospital, Yangzhou
  - Affiliated Hospital, Guangdong Medical College, Zhanjiang
  - Henan Provincial People's Hospital, Zhengzhou
  - Zhengzhou People's Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polverino E, Goeminne PC, McDonnell MJ, Aliberti S, Marshall SE, Loebinger MR, Murris M, Canton R, Torres A, Dimakou K, De Soyza A, Hill AT, Haworth CS, Vendrell M, Ringshausen FC, Subotic D, Wilson R, Vilaro J, Stallberg B, Welte T, Rohde G, Blasi F, Elborn S, Almagro M, Timothy A, Ruddy T, Tonia T, Rigau D, Chalmers JD. European Respiratory Society guidelines for the management of adult bronchiectasis. Eur Respir J. 2017 Sep 9;50(3):1700629. doi: 10.1183/13993003.00629-2017. Print 2017 Sep. PMID 28889110
- [Background] Hill AT, Sullivan AL, Chalmers JD, De Soyza A, Elborn SJ, Floto AR, Grillo L, Gruffydd-Jones K, Harvey A, Haworth CS, Hiscocks E, Hurst JR, Johnson C, Kelleher PW, Bedi P, Payne K, Saleh H, Screaton NJ, Smith M, Tunney M, Whitters D, Wilson R, Loebinger MR. British Thoracic Society Guideline for bronchiectasis in adults. Thorax. 2019 Jan;74(Suppl 1):1-69. doi: 10.1136/thoraxjnl-2018-212463. No abstract available. PMID 30545985
- [Background] Aliberti S, Masefield S, Polverino E, De Soyza A, Loebinger MR, Menendez R, Ringshausen FC, Vendrell M, Powell P, Chalmers JD; EMBARC Study Group. Research priorities in bronchiectasis: a consensus statement from the EMBARC Clinical Research Collaboration. Eur Respir J. 2016 Sep;48(3):632-47. doi: 10.1183/13993003.01888-2015. Epub 2016 Jun 10. PMID 27288031
- [Background] White L, Mirrani G, Grover M, Rollason J, Malin A, Suntharalingam J. Outcomes of Pseudomonas eradication therapy in patients with non-cystic fibrosis bronchiectasis. Respir Med. 2012 Mar;106(3):356-60. doi: 10.1016/j.rmed.2011.11.018. Epub 2011 Dec 26. PMID 22204744
- [Background] Vallieres E, Tumelty K, Tunney MM, Hannah R, Hewitt O, Elborn JS, Downey DG. Efficacy of Pseudomonas aeruginosa eradication regimens in bronchiectasis. Eur Respir J. 2017 Apr 12;49(4):1600851. doi: 10.1183/13993003.00851-2016. Print 2017 Apr. No abstract available. PMID 28404646
- [Background] Blanco-Aparicio M, Saleta Canosa JL, Valino Lopez P, Martin Egana MT, Vidal Garcia I, Montero Martinez C. Eradication of Pseudomonas aeruginosa with inhaled colistin in adults with non-cystic fibrosis bronchiectasis. Chron Respir Dis. 2019 Jan-Dec;16:1479973119872513. doi: 10.1177/1479973119872513. PMID 31480862
- [Background] Orriols R, Hernando R, Ferrer A, Terradas S, Montoro B. Eradication Therapy against Pseudomonas aeruginosa in Non-Cystic Fibrosis Bronchiectasis. Respiration. 2015;90(4):299-305. doi: 10.1159/000438490. Epub 2015 Sep 5. PMID 26340658
- [Background] Pieters A, Bakker M, Hoek RAS, Altenburg J, van Westreenen M, Aerts JGJV, van der Eerden MM. The clinical impact of Pseudomonas aeruginosa eradication in bronchiectasis in a Dutch referral centre. Eur Respir J. 2019 Apr 11;53(4):1802081. doi: 10.1183/13993003.02081-2018. Print 2019 Apr. No abstract available. PMID 30635292